CLINICAL TRIAL: NCT03200847
Title: Pembrolizumab and All-Trans Retinoic Acid in Combination Treatment of Advanced Melanoma
Brief Title: Pembrolizumab and All-Trans Retinoic Acid Combination Treatment of Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1080.cc; PMID 36378549 (Other: PubMed)
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Stage IV Melanoma; Stage III Melanoma; Advanced Melanoma
Keywords: Pembrolizumab; All-Trans Retinoic Acid
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with All-Trans Retinoic Acid (Experimental): Patients will receive pembrolizumab infusions every three weeks. Patients will also receive 3 days of all-trans retinoic acid treatment surrounding each of the first 4 infusions of pembrolizumab, beginning one day prior to the infusion (a total of 12 days of all-trans retinoic acid).
  Interventions: Drug: Pembrolizumab with All-Trans Retinoic Acid

INTERVENTIONS:
Drug: Pembrolizumab with All-Trans Retinoic Acid — All the patients will receive 200mg Q3W pembrolizumab treatment plus the supplemental treatment of 150 mg/m2 All-Trans Retinoic Acid orally for 3 days surrounding each of the first four infusions of pembrolizumab
  Other Names: VESANOID; Keytruda

SUMMARY:
This is a Phase I/Ib investigator-initiated open label of the combination of VESANOID and pembrolizumab treatment.

DETAILED DESCRIPTION:
Primary Objective

* To identify the MTD and RP2D of the combination of pembrolizumab and ATRA.

Secondary Objective:

* Describe the safety and toxicity of combined treatment with pembrolizumab and all-trans retinoic acid (ATRA) [brand name VESANOID] in melanoma patients.
* To assess the anti-tumor activity in terms of a). The reduction in MDSC (immunosuppressive myeloid -derived suppressor cells) frequency and suppressive function (measured as a continuous variable)in peripheral blood of advanced melanoma patients undergoing pembrolizumab and VESANOID combination therapy. b). progression free survival.

Exploratory Objective

* To determine the clinical outcomes with tumor-specific T cell responses.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced melanoma (unresectable Stage III or Stage IV Melanoma).
2. Planned standard treatment with pembrolizumab.
3. Be willing and able to provide written informed consent for the trial.
4. State willingness to comply with all study procedures and be available for the duration of the trial.
5. Be ≥ 18 years of age on day of signing informed consent.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined in Table 1 of the protocol.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential (Section 6.5.2 - Contraception) must be willing to use an adequate method of contraception as outlined in Section 6.5.2 of the protocol - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential (Section 6.5.2- Contraception) must agree to use an adequate method of contraception as outlined in Section 6.5.2 of the protocol - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis).
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Subjects with chronic conditions such as vision changes from plaque radiation therapy for ocular melanoma or prior hearing loss that is not reasonably expected to be exacerbated by the investigational product may be included.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
18. Has known sensitivity to retinoic acid derivatives.
19. Has a medical history of allogenic stem cell transplant or received a solid organ transplant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin McCarter, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobin RP, Cogswell DT, Cates VM, Davis DM, Borgers JSW, Van Gulick RJ, Katsnelson E, Couts KL, Jordan KR, Gao D, Davila E, Medina TM, Lewis KD, Gonzalez R, McFarland RW, Robinson WA, McCarter MD. Targeting MDSC Differentiation Using ATRA: A Phase I/II Clinical Trial Combining Pembrolizumab and All-Trans Retinoic Acid for Metastatic Melanoma. Clin Cancer Res. 2023 Apr 3;29(7):1209-1219. doi: 10.1158/1078-0432.CCR-22-2495. PMID 36378549

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No de-escalation occurred. All subjects received 150 mg/m2 for 3 days before and after each of the first four infusions of pembrolizumab.
Period: Overall Study
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (13.38843)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of Pembrolizumab
Description: MTD is defined as the highest dose level with no more than 3 DLTs reported in 6 DLT-evaluable subjects. A target toxicity rate of approximately 33% of all 24 patients will be used to establish the RP2D. This is one part of the pembrolizumab-ATRA combination treatment.
Time Frame: 21 days from first dose of combined treatment
Population: The analysis population is 24 patients rather than 25 because one patient was not on treatment long enough to be evaluated for any outcomes.
Measure: Number; unit: mg
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 24
mg | 200

2. Secondary Outcome: Number of Patients With a Dose-Limiting Toxicity (DLT) for the Combined Treatment of Pembrolizumab and All-Trans Retinoic Acid
Description: Toxicity is evaluated according to NCI CTCAE Version 4.0. A dose limiting toxicity (DLT) is defined as any grade 3 or higher adverse event related to VESNOID (the all-trans retinoic acid) and/or pembrolizumab.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 24
Participants | 5

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival was calculated from treatment start date to data cutoff date.
Time Frame: up to 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 24
months | 20.3 [7.6 to NA] — The upper limit of the calculated 95% confidence interval was not estimable because there were not enough patients who had events at later timepoints to get a reliable upper estimate.

4. Secondary Outcome: Percent Change in Anti-Tumor Activity
Description: Anti-tumor activity will be determined by the percent change in MDSC (immunosuppressive myeloid-derived suppressor cells) frequency in peripheral blood of advanced melanoma patients undergoing the combined treatment of pembrolizumab and All-Trans Retinoic Acid (ATRA). Pre-treatment levels will be compared to post-treatment levels, where post-treatment means 4-6 weeks after stopping ATRA. MDSCs include CD45+, CD3-, CD19-, CD56-, CD11b+, CD33+, and HLA-DR-/low.
  In the original protocol, suppressive function was included as part of this outcome measure to assess anti-tumor activity. However, this analysis could not be performed because the decrease in concentration of MDSCs after treatment resulted in inadequate data for the planned assays.
Time Frame: Pre-treatment (0-30 days before first ATRA administration) and post-treatment (84-130 days after first ATRA administration)
Population: Percent change in MDSC was computed both in total and separately for i) patients that responded to therapy, and ii) patients that did not respond to therapy. Response was evaluated using RECIST v1.1 criteria. The analysis population for this outcome measure is 23 patients because one patient did not complete a post-treatment blood draw.
Measure: Mean (Standard Deviation); unit: percent change from pre-treatment value
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 23
percent change from pre-treatment value
  Responding patients: number analyzed (Participants) | 17
  Responding patients | -48.6 (54.4)
  Non-responding patients: number analyzed (Participants) | 6
  Non-responding patients | 109.7 (224.6)
  Overall | -7.3 (136.6)

5. Primary Outcome: Maximally Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of All-Trans Retinoic Acid
Description: MTD is defined as the highest dose level with no more than 3 DLT reported in 6 DLT-evaluable subjects. A target toxicity rate of approximately 33% of all 24 patients will be used to establish the RP2D. This dose is one part of the pembrolizumab-ATRA combination treatment.
Time Frame: 21 days from first dose of combined treatment
Population: as for outcome 1
Measure: Number; unit: mg/m2
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
Number analyzed (Participants) | 24
mg/m2 | 150

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pembrolizumab With All-Trans Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab With All-Trans Retinoic Acid (N=25)
Adrenal insufficiency (Renal and urinary disorders) | 1 (1)
DVT (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Encephalopathy (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Shoulder Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Malignant Neoplasm Prostate Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Event (Nervous system disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Blood and lymphatic system disorders) | 1 (1)
Intramedullary nail fixation of L humerus surgery (Surgical and medical procedures) | 1 (1)
Thrombolytic Event (Blood and lymphatic system disorders) | 1 (1)
Acute kidney insufficiency (Renal and urinary disorders) | 1 (1)
Altered mental status due to new brain mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab With All-Trans Retinoic Acid (N=25)
Abdominal Pain (General disorders) | 3 (3)
Adrenal Insufficiency (Endocrine disorders) | 2 (2)
Alanine aminotransferase increased (Gastrointestinal disorders) | 6 (8)
Alkaline Phosphatase Increase (Blood and lymphatic system disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (8)
anorexia (General disorders) | 2 (2)
anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (General disorders) | 2 (3)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 5 (5)
Back Pain (General disorders) | 3 (3)
Bladder Infection (Infections and infestations) | 1 (2)
Hypothyroid (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Elevated TSH (Endocrine disorders) | 1 (1)
Chronic anticoagulation (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (3)
R Bundle Branch Block w/L Anterior Fascia Block (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (General disorders) | 6 (7)
Creatinine Increased (Renal and urinary disorders) | 4 (4)
Dehydration (General disorders) | 2 (2)
Dental Caries (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Dizziness (General disorders) | 5 (5)
Dry Mouth (General disorders) | 5 (5)
Dry Skin (General disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Ear Wound (Ear and labyrinth disorders) | 1 (1)
Ear pain (General disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 3 (3)
Endocrine Disorders (Endocrine disorders) | 2 (2)
epistaxis (General disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Sore Eyes (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 16 (28)
Fever (Infections and infestations) | 2 (2)
Flank Pain (General disorders) | 1 (1)
Flu like Symptoms (General disorders) | 1 (1)
Flushing (Cardiac disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 3 (4)
Small Bowel obstruction (Gastrointestinal disorders) | 1 (1)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1)
Nausea without Vomiting (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Sinus Congestion (General disorders) | 1 (1)
Reduced Stamina (General disorders) | 1 (1)
Decreased Appetite (General disorders) | 3 (3)
Night Sweats (General disorders) | 1 (1)
Runny Nose (General disorders) | 1 (2)
Dry lips (General disorders) | 1 (1)
Elevated PSA (Renal and urinary disorders) | 1 (1)
Pneumomesentery (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 20 (46)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoids (General disorders) | 1 (1)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1)
Portal Vein/Hepatic Thrombosis (Hepatobiliary disorders) | 1 (1)
LFT Elevation (Hepatobiliary disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (2)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (2)
Hyperglycemia (Endocrine disorders) | 2 (2)
Hypoalbuminemia (Vascular disorders) | 1 (1)
Hypokalemia (Gastrointestinal disorders) | 2 (3)
Hyponatremia (General disorders) | 1 (3)
Hypotension (Cardiac disorders) | 1 (2)
COVID-19 (Infections and infestations) | 3 (3)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (General disorders) | 2 (2)
Intracranial Hemorrhage (General disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Libido decreased (General disorders) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 2 (2)
Diabetes mellitus Type II (Metabolism and nutrition disorders) | 1 (1)
Loss of Weight (Metabolism and nutrition disorders) | 3 (3)
Oral Mucositis (Skin and subcutaneous tissue disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Left Inguinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Tightness (Musculoskeletal and connective tissue disorders) | 2 (5)
Chest Tingles (Musculoskeletal and connective tissue disorders) | 1 (1)
Penis Tingles (Musculoskeletal and connective tissue disorders) | 1 (1)
Soreness in Penis (Metabolism and nutrition disorders) | 1 (1)
Right Upper Quadrant Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia Rheumatica Symptoms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (General disorders) | 8 (15)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Osteoporsis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Palipations (Cardiac disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Photosensitivity (Eye disorders) | 1 (1)
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 (5)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Forgetfulness (Psychiatric disorders) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 7 (11)
Enlarged Prostate (Renal and urinary disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scrotal Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Dry desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Generalized Itchy Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Left Chest Papule of Unknown Origin (Skin and subcutaneous tissue disorders) | 1 (1)
Xerosis over BUE (Skin and subcutaneous tissue disorders) | 1 (1)
Tinea Pedis - Bilateral (Skin and subcutaneous tissue disorders) | 1 (1)
pruritis on Abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Desquamation - Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Fingers Peeling (Skin and subcutaneous tissue disorders) | 1 (1)
Erythematous Rash on Trunk (Skin and subcutaneous tissue disorders) | 1 (1)
Erythematous Rash on Back (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar/plantar xeroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Post-Operative Dental Pain (Surgical and medical procedures) | 1 (1)
Tinnituts (General disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Upper Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary Tract infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (9)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (3)
Acute urinary Retention (Renal and urinary disorders) | 1 (1)
Right Eye Stye (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03200847/Prot_SAP_ICF_000.pdf